CLINICAL TRIAL: NCT04079478
Title: The AID Study: Artificial Intelligence for Colorectal Adenoma Detection
Acronym: AID
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2363
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer
Keywords: Artificial Intelligence
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI: Artificial Intelligence colonoscopy
  Interventions: Other: AI
- Control: White light colonoscopy

INTERVENTIONS:
Other: AI — Artificial intellignece colonoscopy
  Groups: AI

SUMMARY:
Colonoscopy is clinically used as the gold standard for detection of colon cancer (CRC) and removal of adenomatous polyps. Despite the success of colonoscopy in reducing cancer-related deaths, there exists a disappointing level of adenomas missed at colonoscopy. "Back-to-back" colonoscopies have indicated significant miss rates of 27% for small adenomas (< 5 mm) and 6% for adenomas of more than 10 mm in diameter. Studies performing both CT colonography and colonoscopy estimate that the colonoscopy miss rate for polyps over 10 mm in size may be as high as 12%. The clinical importance of missed lesions should be emphasized because these lesions may ultimately progress to CRC8.

Limitations in human visual perception and other human biases such as fatigue, distraction, level of alertness during examination increases such recognition errors and way of mitigating them may be the key to improve polyp detection and further reduction in mortality from CRC. In the past years, a number of CAD systems for detection of polyps from endoscopy images have been described. However, the benefits of traditional CAD technologies in colonoscopy appear to be contradictory, therefore they should be improved to be ultimately considered useful. Recent advances in artificial intelligence (AI), deep learning (DL), and computer vision have shown potential to assist polyp detection during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

All 40-80 years-old subjects undergoing a colonoscopy.

Exclusion Criteria:

* subjects with personal history of CRC, or IBD.
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale > 2 in any colonic segment).
* patients with previous colonic resection.
* patients on antithrombotic therapy, precluding polyp resection.
* patients who were not able or refused to give informed written consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the observed prevalence of adenomas (35%) among patients undergoing colonoscopies at our center within the last 12 months, a sample size of 322 subjects per arm could allow for a 90% power to show the non-inferiority (primary end-point) of the AI-aided arm by excluding that the one-side 95% CI will exclude a difference of 10% in favour of the standard group. Such sample size will also have a 80% power to detect as statistical significant (α=0.05; two-sided test) a 10% absolute increase in the detection rate of adenomas in the AI-aided arm (secondary end-point).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Additional diagnostic yield obtained by AI-aided colonoscopy to the yield obtained by the Standard (high-definition) colonoscopy | 3 Months
  To compare the additional diagnostic yield obtained by AI-aided colonoscopy to the yield obtained by the Standard (high-definition) colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No